CLINICAL TRIAL: NCT04690725
Title: Phase I Study of TQB3525, Phosphatidylinositol-3-Kinase α and δ Inhibitors, in Patients With Advanced Bone Sarcomas
Brief Title: TQB3525 for Advanced Bone Sarcomas With PI3KA Mutations or PTEN Loss
Acronym: TQBSP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Director, Head of Msculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma12
Record Dates: First submitted 2020-12-25; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Safety Issues; Efficacy, Self
Keywords: osteosarcoma; ewing sarcoma; chondrosarcoma; PI3KA mutation; PTEN loss; TQB3525
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Chondrosarcoma | interventions — TQ-B3525

STUDY DESIGN:
Intervention Model Description: TQB3525 orally taken
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3525 arm (Experimental): 3+3 design for phase I for RP2D (Recommended Phase 2 Dose) for adolescents (12-17 years old) (15mg QD or 20mg QD); phase II for efficacy exploration for another 17 patients using RP2D QD
  Interventions: Drug: TQB3525

INTERVENTIONS:
Drug: TQB3525 — TQB3525 is an orally bioavailable, potent, class I kinase inhibitors of PI3Ka and PI3Kd.

SUMMARY:
The PI3K, protein kinase B (AKT), and mTOR signaling network promotes cell growth, survival, metabolism, and motility, but becomes a critical oncogenic driver under aberrant conditions that control the tumor microenvironment and angiogenesis. The PI3K-AKT-mTOR axis is the most frequently deregulated signaling pathway in primary osteosarcoma and other bone tumors. PI3Ka has high rates of 25-50% activating mutations associated with tumor formation in osteosarcoma. Other causes of pathway hyperactivation include loss of function of the tumor suppressor PTEN, gain-of-function mutations in AKT and PDK1, or upregulation of receptor tyrosine kinases. TQB3525 is an orally bioavailable, potent, dual catalytic site inhibitor of PI3Ka and PI3Kd. Tumor growth inhibition has been demonstrated in multiple xenograft osteosarcoma models with PI3K-mutant, PTEN-null cell lines. The investigators try to investigate TQB3525 in primary osteosarcoma and other bone tumors for its safety, tolerability, dose-limiting toxicities (DLT), MTD and antitumor efficacy.

ELIGIBILITY:
Inclusion Criteria:

* progression upon first-line chemotherapy;
* with target lesions according to RECIST 1.1;
* geno-profiling with PI3KA mutations or PTEN loss;
* ECOG PS status 0 or 1 with a life expectancy >3 months;
* adequate renal, hepatic, and hematopoietic function;

Exclusion Criteria:

* been previously exposed to other TKIs;
* had central nervous system metastasis;
* had other kinds of malignant tumors at the same time;
* had cardiac insufficiency or arrhythmia;
* had uncontrolled complications such as diabetes mellitus, coagulation disorders, urine protein ≥ ++, and so on;
* had pleural or peritoneal effusion that needed to be handled by surgical treatment;
* had other infections or wounds;
* pregnant or breastfeeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
toxicity profiles | 6 months
  according to CTCAE 5.0

SECONDARY OUTCOMES:
progression free survival | 6 months
  from starting treatment to progression/death
overall survival | 2 years
  from starting treatment to death

OTHER OUTCOMES:
fasting triglyceride | 6 months
  dynamic changes from Peripheral Blood
fasting lipoprotein | 6 months
  dynamic changes from Peripheral Blood
fasting insulin | 6 months
  dynamic changes from Peripheral Blood

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Ph.D and M.D., Principal Investigator — Chinese Sarcoma Study Group
Locations (1):
- Peking University Shougang Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No